CLINICAL TRIAL: NCT02726815
Title: Pain and Symptoms in Children With Advanced Cancer: a Longitudinal Study to Develop a Comprehensive Symptom Inventory
Brief Title: Developing a Symptom List for Children With Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4385
Record Dates: First submitted 2016-03-22; First posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Paediatric Oncology Palliative Care
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire based study using a symptom assessment tool

SUMMARY:
Primary Objective

The aim of this research study is to develop a comprehensive inventory of symptoms that occur in children with advanced cancer who are receiving a specialist palliative care service.

Secondary Objectives

* To assess correlation between parent, child and nurse scores on the Memorial Symptom Assessment Scale (MSAS).
* To identify symptom prevalence in children with advanced cancer as identified by the child/young person (CYP), nurse and parent (to be analysed separately for parent, child and nurse).
* To identify whether there are any symptoms missing from the age appropriate MSAS as identified by the CYP, nurse and parent (to be analysed separately for parent, child and nurse).
* To identify whether any items on the age appropriate MSAS are not relevant to the population being studied (to be analysed separately for parent, child and nurse).
* To identify which symptoms cause the most distress as identified by the CYP, nurse and parent (to be analysed separately for parent, child and nurse).
* To identify degree of severity of each symptom as identified by the CYP, nurse and parent (to be analysed separately for parent, child and nurse).
* To identify which symptoms occur most frequently as identified by the CYP, nurse and parent (to be analysed separately for parent, child and nurse).
* To assess the trends between phase of illness and symptom profile, severity and distress.

ELIGIBILITY:
Inclusion Criteria:

* Any child/young person (CYP) aged 7 to 17 years and 364 days referred and accepted to the palliative care service (PATCH team) at the Royal Marsden (RM) will be eligible for inclusion. The PATCH team is responsible for co-ordinating palliative care services for children with both malignant and non-malignant conditions in the South Thames and South East Coast areas. The team can provide home visits, local hospital and hospice visits for symptom and palliative care advice. The team are also available by telephone 24 hours a day, 365 days a year to provide symptom advice to families and health care professionals from all settings who are caring for children known to the team. Acceptance to this service is via multidisciplinary team (MDT) discussion.

Exclusion Criteria:

* Severe cognitive impairment in the parent/carer
* Lack of fluent English
* Lack of ability to read and write English
* Psychological concerns about the CYP and/or parent/carer. All potential participants will be discussed with the psychosocial team before being invited to participate.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any child/young person (CYP) aged 7 to 17 years and 364 days referred and accepted to the paediatric symptom care teams at the Royal Marsden will be eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of all symptoms identified by child using the age appropriate Memorial Symptom Assessment Scale. | 18 months
Prevalence of all symptoms identified by the parent using the same assessment tool as the child | 18 months
Prevalence of all symptoms identified by the nurse | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Karenia Anderson, MbchB, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Plan to share internally at meetings as well as at conferences. Also plan to submit for publication in a peer reviewed journal.